CLINICAL TRIAL: NCT02489526
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injections for Post-Operative Pain Following Laparoscopic Colorectal Surgery
Brief Title: Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injections for Post-Operative Pain Following Colorectal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVZ149-POP-P2-US001
Record Dates: First submitted 2015-06-18; First posted 2015-07-03 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2019-03

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VVZ-149 Injections (Experimental)
  Interventions: Drug: VVZ-149 Injections
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 Injections — Experimental group will receive a loading dose of 1.8 mg/kg VVZ-149 intravenous infusion for 0.5 hour followed by a maintenance dose of 1.3 mg/kg/h VVZ-149 intravenous infusion for 7.5 hours.
  Other Names: Opiranserin Injections
  Arms: VVZ-149 Injections
Drug: Placebo — Placebo group will receive the corresponding amount of placebo.
  Arms: Placebo

SUMMARY:
The purpose of this Phase 2 study is to evaluate the efficacy and safety of an analgesic drug candidate, VVZ-149 Injections. The study is designed as randomized, double-blind, parallel, placebo-controlled study.

DETAILED DESCRIPTION:
VVZ-149 is a dual antagonist of GlyT2 and 5HT2A. GlyT2 blockage increases inhibitory synaptic transmission by glycine in the spinal cord, resulting in a reduction of pain transmissions to the brain. 5HT2A blockage decreases descending serotonergic facilitatory modulation on pain transmission by the brain and reduces nociceptor activation in peripheral nerves, which are primary sources of pain in post-surgical pain. VVZ-149 has been shown to have comparable efficacy to morphine in well controlled (blind, complete randomization with a positive control) animal studies using rat models of post-operative pain and formalin-induced pain. The PK/PD study in animals indicates that therapeutic plasma concentration in human subjects will be 600-1,900 ng/ml. A clinical Phase 1 study performed in healthy subjects has shown no clinically significant adverse events up to a plasma concentration level of 3,261 ng/ml other than brief symptoms of mild nausea or dizziness, and mild somnolence when the plasma exposure level is more than 2,000 ng/ml.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age between 18-70, inclusive.
2. Pain intensity (NRS) ≥4 at initial post-operative measurement in PACU.
3. Subjects undergoing planned laparoscopic colorectal surgery.
4. Ability to provide written informed consent.
5. Ability to understand study procedures and communicate clearly with the investigator and staff.
6. American Society of Anesthesiologists (ASA) risk class of I to III.

Exclusion Criteria:

< Surgical Factors >

1. Emergency or unplanned surgery.
2. Repeat operation (e.g., previous surgery within 30 days for same condition).
3. Cancer-related condition causing preoperative pain in site of surgery.

   < Subject Characteristics >
4. Women with childbearing potential (Women age 18-55 must undergo pregnancy test).
5. Women who are pregnant or breastfeeding.
6. Chronic pain diagnosis (e.g., ongoing pain at baseline with NRS ≥ 4/10).
7. Unstable or poorly controlled psychiatric condition (e.g., untreated PTSD, anxiety, or depression) Subjects who take stable doses (same dose >30 days) of antidepressants and anti-anxiety drugs may be included.
8. Unstable or acute medical condition (e.g., unstable angina, congestive heart failure, renal failure, hepatic failure, AIDS).

   < Drug, Alcohol, and Pharmacological Considerations >
9. Renal or hepatic impairment.
10. History of alcohol, opiate or other drug abuse or dependence within 12 months prior to Screening (TICS alcohol/drug screen will be performed at Screening).
11. Ongoing or recent (within 30 days prior to surgery) use of steroids, opioids, or antipsychotics.
12. Alcohol consumption within 24 hours of surgery.
13. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) or acetaminophen within 24 hours of surgery.
14. Use of herbal agents or nutraceuticals (i.e., chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian) within 7 days prior to surgery.

    < Anesthetic and Other Exclusion Considerations >
15. Use of neuraxial or regional anesthesia related to the surgery.
16. Use of local anesthetic wound infiltration > 20 ml of 1% lidocaine
17. Use of ketamine, gabapentin, pregabalin, or lidocaine (>1 mg/kg) intra or peri-operatively, or within 24 hours of surgery.
18. Subjects with known allergies to hydromorphone.
19. Subjects who received another investigational drug within 30 days of scheduled surgery.
20. Subjects who have long PR (>200 msec) or prolonged QTc (> 450 msec) at Screening or on an EKG done immediately prior to dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Difference over 8-hours post-dose (SPID8) | 8 hours post-dose
  SPID8 using Numerical Pain Rating Scale (NRS, 0-10) measured up to 8 hours post-dose

SECONDARY OUTCOMES:
Difference of Opioid Consumption between Study Groups | 0-2, 2-4, 4-6, 6-8, 8-12, 12-16, and 16-24 hours post-dose
Change of Pain Intensity (NRS) | 9 and 24 hours post-dose
Change of Pain Relief (PR) assessed using a 6-point categorical scale | 9 and 24 hours post-dose
Comparison of Global Measurement of Subject Satisfaction between Study Groups | 8 and 24 hours post-dose
Change of Richmond Agitation-Sedation Scale | 9 and 24 hours post-dose
Change of Incidence of Postoperative Nausea and Vomiting | 8 and 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Nedeljkovic SS, Song I, Bao X, Zeballos JL, Correll DJ, Zhang Y, Ledley JS, Bhandari A, Bai X, Lee SR, Cho S. Exploratory study of VVZ-149, a novel analgesic molecule, in the affective component of acute postoperative pain after laparoscopic colorectal surgery. J Clin Anesth. 2022 Feb;76:110576. doi: 10.1016/j.jclinane.2021.110576. Epub 2021 Nov 15. PMID 34794108
- [Derived] Song I, Cho S, Nedeljkovic SS, Lee SR, Lee C, Kim J, Bai SJ. Role of VVZ-149, a Novel Analgesic Molecule, in the Affective Component of Pain: Results from an Exploratory Proof-of-Concept Study of Postoperative Pain following Laparoscopic and Robotic-Laparoscopic Gastrectomy. Pain Med. 2021 Sep 8;22(9):2037-2049. doi: 10.1093/pm/pnab066. PMID 33624798
- [Derived] Nedeljkovic SS, Correll DJ, Bao X, Zamor N, Zeballos JL, Zhang Y, Young MJ, Ledley J, Sorace J, Eng K, Hamsher CP, Maniam R, Chin JW, Tsui B, Cho S, Lee DH. Randomised, double-blind, parallel group, placebo-controlled study to evaluate the analgesic efficacy and safety of VVZ-149 injections for postoperative pain following laparoscopic colorectal surgery. BMJ Open. 2017 Feb 17;7(2):e011035. doi: 10.1136/bmjopen-2016-011035. PMID 28213593